CLINICAL TRIAL: NCT02466984
Title: Subcutaneous Route and Pharmacology of Metoclopramide
Acronym: SOPHA-Méto
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2014/10
Record Dates: First submitted 2015-05-29; First posted 2015-06-09 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Nausea; Vomiting
Keywords: metoclopramide; subcutaneous route; palliative care; pharmacology; bioavailability; nausea; vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metoclopramide subcutaneous (Experimental): every two days, first from 10 to 20 and then from 20 to 30 mg/d
  Interventions: Drug: metoclopramide intravenous
- metoclopramide intravenous (Active Comparator): first from 10 to 20 and then from 20 to 30 mg/d
  Interventions: Drug: metoclopramide intravenous

INTERVENTIONS:
Drug: metoclopramide intravenous — Administration route
  Other Names: Primperan

SUMMARY:
Subcutaneous (SC) route has become a standard of care of many drugs administration in palliative medicine. A preliminary study showed that, although it was widely adopted among palliative care practitioners for routinely prescribed medications, standards of proof are still lacking for many molecules. Among them, metoclopramide is a largely employed drug for nausea and vomiting treatment, particularly in palliative care and oncology. Therefore, the investigator aim to study absorption and efficacy of subcutaneous administration of metoclopramide.

DETAILED DESCRIPTION:
In this cross-over study, each patient receives subcutaneous and intravenous metoclopramide, with a randomized order of administration. During each perfusion phases, metoclopramide is administrated with continuous flow, doses being increased every two days, first from 10 to 20 and then from 20 to 30 mg/d. In order to guarantee plasmatic balance during route change, the first dose of the second phase is extended for three days. Metoclopramide plasmatic concentration is measured at inclusion and at the end of each dose administration, with a total of 7 dosages.

Principal purpose of this research is to clarify subcutaneous bioavailability of metoclopramide. For this meaning, the mean difference between all subcutaneous and intravenous concentration ratios is compared. Secondary purposes consist of: calculating metoclopramide subcutaneous bioavailability for each study dose (10, 20 and 30 mg/d); describing dose-bioavailability relation for subcutaneous metoclopramide; comparing dose-concentration relationship of intravenous and subcutaneous metoclopramide; studying local tolerance by checking all inflammatory signs surrounding injection site; evaluating clinical efficacy by comparing between the two groups the number of vomiting episodes, use of Serotonin receptor antagonists and the nausea scores on a 11-level numerical scale.

Eighteen patients have to be analysed at least. For each patient not having completed the study, one more will be included in order to reach the eighteen necessary patients. Therefore, it is expected to include twenty-four patients. Included population characteristics will be described. A three-dimensional analysis with period, subject and dose is performed to determine metoclopramide absolute bioavailability. For secondary criteria, dose-concentration relation is analysed with a four-dimensional analysis; dose-bioavailability and dose-concentration relations are described by linear and log-linear regression. For principal purpose, only results of patients having completed the study are part of this aforementioned analyse.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years
* Patients hospitalized at the palliative medical care unit of University Hospital Bordeaux
* Patient whose life expectancy is greater to 4 weeks
* Patients suffering from nausea the day of inclusion with a greater than or equal score to 3/10 on a numerical scale (FR) from 0 to 10 and / or have had at least one vomiting within three days prior to inclusion
* Patients may be infused through an IV and subcutaneous (SC)
* Patient can communicate verbally or in writing
* Patients affiliates or beneficiaries of a social security fund
* Patient has given his written consent

Exclusion criteria

* Pregnant or breastfeeding women
* Current Treatment for severe and progressive threatening disease
* Treatment with oral or injectable metoclopramide within 3 days prior to inclusion
* Treatment with levodopa or dopamine agonists in progress
* Neuroleptic Processing
* Patient with lesion occlusive syndrome
* Patients at risk of gastrointestinal perforation
* Patient with clinical signs of gastrointestinal bleeding
* Parkinson's disease
* Patients with epilepsy not controlled by anti-seizure treatment
* Patients suffering from liver failure
* Patients with a heart rate less than 60 beats / min at baseline
* Patients with systolic blood pressure less than or equal to 90 mmHg at baseline
* History of allergy to metoclopramide
* History of allergy to ondansetron
* Previous history of tardive dyskinesia to neuroleptics or metoclopramide
* Previous history of pheochromocytoma
* Previous history of methemoglobinemia with metoclopramide
* History of deficit NADH-cytochrome b5 reductase
* Patient deprived of liberty by judicial or administrative decision
* Major protected by law
* Exclusion period Patient relative over another protocol.

Exclusion criteria

* Pregnant woman (blood β-HCG dosage ≥ 5 IU / L)
* Patients with a creatinine clearance less than or equal to 60 mL / min at baseline
* Patient with cardiac conduction disorders on ECG
* Patients with electrolyte imbalance in electrolytes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of SubCutaneus administration metoclopramide | 13 days
  Calculated by the average ratio of plasma concentrations between SC route and IV on all doses of the study (10, 20 and 30 mg / d)

SECONDARY OUTCOMES:
Absolute bioavailability of metoclopramide subcutaneously at each dose of the study (10, 20 and 30 mg / d) | 13 days
  Calculated by the ratio of plasma concentrations between SC route and the IV route;
Dose-bioavailability of metoclopramide for the SC route | 13 days
Relations plasma concentration-dose metoclopramide subcutaneously and intravenously | 13 days
  Measured through their apparent clearances
Cutaneous inflammatory signs and subcutaneous at the puncture site | During 13 days
Numeric scale ranging from 0 to 10 for nausea | During 13 days
Number of vomiting in the dose level; | During 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu FRASCA, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux - St André, Bordeaux, Aquitaine, France